CLINICAL TRIAL: NCT01960933
Title: Primary PCI in Patients With ST-elevation Myocardial Infarction and Multivessel Disease: Treatment of Culprit Lesion Only or Complete Revascularization (DANAMI-3-PRIMULTI) A Randomised Comparison of the Clinical Outcome After Complete Revascularisation Versus Treatment of the Infarct-related Artery Only During Primary Percutaneous Coronary Intervention
Brief Title: Primary PCI in Patients With ST-elevation Myocardial Infarction and Multivessel Disease: Treatment of Culprit Lesion Only or Complete Revascularization
Acronym: PRIMULTI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Engstrom, MD, Senior Consultant, DMSCi, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DANAMI-3-PRIMULTI
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: ST-elevation Myocardial Infarction; Multi Vessel Disease
Keywords: STEMI; MVD; Full revascularization; Culprit lesion revascularization only; Primary PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Culprit lesion revascularization (Active Comparator): Only the culprit lesion is treated whereas other study lesions are left un-treated.
  Interventions: Procedure: Percutaneous coronary intervention
- Full revascularization (Active Comparator): Culprit lesion is treated initially and all other lesions with diameter stenosis angiographically >50% and FFR <0.80 are treated in a separate procedure within the index hospitalization. Stenoses > 90% are treated without prior FFR.
  Interventions: Procedure: Percutaneous coronary intervention; Procedure: FFR

INTERVENTIONS:
Procedure: Percutaneous coronary intervention
Procedure: FFR
  Arms: Full revascularization

SUMMARY:
In patients with ST-elevation myocardial infarction (STEMI) the primary treatment is acute angioplasty of the acute occlusion (culprit lesion). In STEMI patients with multi vessel disease (MVD) no evidence based treatment of the non-culprit lesions exists. We aim to provide evidence as to whether full revascularization or revascularization of the culprit lesion only provides the best prognosis for the patient.

DETAILED DESCRIPTION:
STEMI patients with MVD (30% of total STEMI population) are - following successful primary angioplasty - randomized to either no additional percutaneous coronary intervention (PCI) of other lesions or full revascularisation guided by fractional flow reserve (FFR).

Eligible coronary arteries must be >2.0 mm in diameter and at the discretion of the operator suitable for PCI. Only arteries with angiographically stenoses > 50% can be randomized. All randomized lesions with diameter stenosis > 50% and < 90% are evaluated by FFR and a FFR value < 0.80 is considered significant and treated. Stenoses >90% are treated without prior FFR.

Full revascularization is a priori obtained by means of PCI. If, however, PCI is considered inferior to coronary artery bypass grafting the latter option can be chosen.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Acute onset of chest pain of < 12 hours' duration.
* ST-segment elevation ≥ 0.1 millivolt in ≥ 2 contiguous leads, signs of a true posterior infarction or documented newly developed left bundle branch block.
* Culprit lesion in a major native vessel.
* MVD (non-culprit vessels with angiographic stenosis >50%)
* Successful primary PCI

Exclusion Criteria:

* Pregnancy.
* Known intolerance of acetylsalicylic acid, clopidogrel, heparin or contrast.
* Inability to understand information or to provide informed consent.
* Haemorrhagic diathesis or known coagulopathy.
* Stent thrombosis
* Significant left main stem stenosis
* Cardiogenic shock at admittance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2011-05; Primary Completion 2015-02 (Actual); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
All cause death, myocardial infarction or revascularization | 1 year
  Composite of all cause mortality, myocardial infarction, or ischemia (either subjective or objective) driven revascularization of non-culprit coronary lesions eligible for and randomized to either of the two treatment arms at the time of the index procedure

SECONDARY OUTCOMES:
Cardiac death or myocardial infarction | 1 year
Hospitalization for acute coronary syndrome or acute heart failure | 1 year
Angina status and quality of life | 1 year
Infarct size in relation to area at risk as determined by MRI | 3 months
Cardiac death, myocardial infarction, repeat revascularisation or occurrence of definite stent thrombosis (according to ARC definition) of non culprit lesions | 2 years
Wall motion index (WMI) determined by echocardiography | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Helqvist, MD, DMSci, Study Chair — Rigshospitalet, Denmark; Thomas Engstrøm, MD, DMSci, Principal Investigator — Rigshospitalet, Denmark; Henning Kelbæk, MD. DMSci, Principal Investigator — Rigshospitalet, Denmark; Lars Køber, MD, Prof., DMSci, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, University of Copenhagen, Copenhagen

REFERENCES:
- [Derived] Elezi B, Marquard JM, Kelbaek H, Nepper-Christensen L, Ahtarovski K, Kyhl K, Goransson C, Islam U, Kober L, Hofsten D, Pedersen F, Vejlstrup NG, Holmvang L, Engstrom T, Lonborg JT. Ten-year prognostic impact of cardiac magnetic resonance endpoints in patients with ST-segment elevation myocardial infarction. Eur Heart J Cardiovasc Imaging. 2026 Jan 6:jeag001. doi: 10.1093/ehjci/jeag001. Online ahead of print. PMID 41493904
- [Derived] Ozbek BT, Islam U, Marquard JM, Kelbaek H, Kunkel JB, Holmvang L, Tilsted HH, Pedersen F, Koeber L, Hofsten D, Eftekhari A, Raungaard B, Bottker HE, Terkelsen CJ, Christiansen E, Khalek IMA, Jensen LO, Engstrom T, Lonborg JT. Ten-year target lesion failure in patients treated with primary PCI: results from DANAMI-3. Open Heart. 2025 Nov 13;12(2):e003588. doi: 10.1136/openhrt-2025-003588. PMID 41238348
- [Derived] Marquard JM, Beske RP, Kelbaek H, Holmvang L, Pedersen F, Clemmensen P, De Backer O, Raungaard B, Eftekhari A, Islam U, Kober L, Tilsted HH, Glinge C, Jabbari R, Scheike T, Hofsten DE, Lonborg JT, Engstrom T. 10-Year Outcome of Complete or Infarct Artery-Only Revascularization in STEMI With Multivessel Disease: The DANAMI-3-PRIMULTI Study. J Am Coll Cardiol. 2025 Jul 15;86(2):119-129. doi: 10.1016/j.jacc.2025.05.013. Epub 2025 May 20. PMID 40392668
- [Derived] Mazhar J, Ekstrom K, Kozor R, Grieve SM, Nepper-Christensen L, Ahtarovski KA, Kelbaek H, Hofsten DE, Kober L, Vejlstrup N, Vernon ST, Engstrom T, Lonborg J, Figtree GA. Cardiovascular magnetic resonance characteristics and clinical outcomes of patients with ST-elevation myocardial infarction and no standard modifiable risk factors-A DANAMI-3 substudy. Front Cardiovasc Med. 2022 Aug 3;9:945815. doi: 10.3389/fcvm.2022.945815. eCollection 2022. PMID 35990971
- [Derived] Ekstrom K, Nielsen JVW, Nepper-Christensen L, Ahtarovski KA, Kyhl K, Goransson C, Bertelsen L, Ghotbi AA, Kelbaek H, Hofsten DE, Kober L, Schoos MM, Vejlstrup N, Lonborg J, Engstrom T. Ischemia From Nonculprit Stenoses Is Not Associated With Reduced Culprit Infarct Size in Patients with ST-Segment-Elevation Myocardial Infarction. Circ Cardiovasc Imaging. 2021 May;14(5):e012290. doi: 10.1161/CIRCIMAGING.120.012290. Epub 2021 May 5. PMID 33951923
- [Derived] Ekstrom K, Nepper-Christensen L, Ahtarovski KA, Kyhl K, Goransson C, Bertelsen L, Ghotbi AA, Kelbaek H, Helqvist S, Hofsten DE, Kober L, Schoos MM, Vejlstrup N, Lonborg J, Engstrom T. Impact of Multiple Myocardial Scars Detected by CMR in Patients Following STEMI. JACC Cardiovasc Imaging. 2019 Nov;12(11 Pt 1):2168-2178. doi: 10.1016/j.jcmg.2019.01.032. Epub 2019 Apr 17. PMID 31005537
- [Derived] Wang LJ, Han S, Zhang XH, Jin YZ. Fractional flow reserve-guided complete revascularization versus culprit-only revascularization in acute ST-segment elevation myocardial infarction and multi-vessel disease patients: a meta-analysis and systematic review. BMC Cardiovasc Disord. 2019 Mar 1;19(1):49. doi: 10.1186/s12872-019-1022-6. PMID 30823897
- [Derived] Nepper-Christensen L, Lonborg J, Hofsten DE, Ahtarovski KA, Bang LE, Helqvist S, Kyhl K, Kober L, Kelbaek H, Vejlstrup N, Holmvang L, Engstrom T. Benefit From Reperfusion With Primary Percutaneous Coronary Intervention Beyond 12 Hours of Symptom Duration in Patients With ST-Segment-Elevation Myocardial Infarction. Circ Cardiovasc Interv. 2018 Sep;11(9):e006842. doi: 10.1161/CIRCINTERVENTIONS.118.006842. PMID 30354595
- [Derived] Kobayashi Y, Lonborg J, Jong A, Nishi T, De Bruyne B, Hofsten DE, Kelbaek H, Layland J, Nam CW, Pijls NHJ, Tonino PAL, Warnoe J, Oldroyd KG, Berry C, Engstrom T, Fearon WF; DANAMI-3-PRIMULTI, FAME, and FAMOUS-NSTEMI Study Investigators. Prognostic Value of the Residual SYNTAX Score After Functionally Complete Revascularization in ACS. J Am Coll Cardiol. 2018 Sep 18;72(12):1321-1329. doi: 10.1016/j.jacc.2018.06.069. PMID 30213322
- [Derived] Falkentoft AC, Rorth R, Iversen K, Hofsten DE, Kelbaek H, Holmvang L, Frydland M, Schoos MM, Helqvist S, Axelsson A, Clemmensen P, Jorgensen E, Saunamaki K, Tilsted HH, Pedersen F, Torp-Pedersen C, Kofoed KF, Goetze JP, Engstrom T, Kober L. MR-proADM as a Prognostic Marker in Patients With ST-Segment-Elevation Myocardial Infarction-DANAMI-3 (a Danish Study of Optimal Acute Treatment of Patients With STEMI) Substudy. J Am Heart Assoc. 2018 May 18;7(11):e008123. doi: 10.1161/JAHA.117.008123. PMID 29776961
- [Derived] Lonborg J, Engstrom T, Kelbaek H, Helqvist S, Klovgaard L, Holmvang L, Pedersen F, Jorgensen E, Saunamaki K, Clemmensen P, De Backer O, Ravkilde J, Tilsted HH, Villadsen AB, Aaroe J, Jensen SE, Raungaard B, Kober L, Hofsten DE; DANAMI 3-PRIMULTI Investigators. Fractional Flow Reserve-Guided Complete Revascularization Improves the Prognosis in Patients With ST-Segment-Elevation Myocardial Infarction and Severe Nonculprit Disease: A DANAMI 3-PRIMULTI Substudy (Primary PCI in Patients With ST-Elevation Myocardial Infarction and Multivessel Disease: Treatment of Culprit Lesion Only or Complete Revascularization). Circ Cardiovasc Interv. 2017 Apr;10(4):e004460. doi: 10.1161/CIRCINTERVENTIONS.116.004460. PMID 28404623
- [Derived] Engstrom T, Kelbaek H, Helqvist S, Hofsten DE, Klovgaard L, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, Clemmensen P, De Backer O, Ravkilde J, Tilsted HH, Villadsen AB, Aaroe J, Jensen SE, Raungaard B, Kober L; DANAMI-3-PRIMULTI Investigators. Complete revascularisation versus treatment of the culprit lesion only in patients with ST-segment elevation myocardial infarction and multivessel disease (DANAMI-3-PRIMULTI): an open-label, randomised controlled trial. Lancet. 2015 Aug 15;386(9994):665-71. doi: 10.1016/s0140-6736(15)60648-1. PMID 26347918
- [Derived] Hofsten DE, Kelbaek H, Helqvist S, Klovgaard L, Holmvang L, Clemmensen P, Torp-Pedersen C, Tilsted HH, Botker HE, Jensen LO, Kober L, Engstrom T; DANAMI 3 Investigators. The Third DANish Study of Optimal Acute Treatment of Patients with ST-segment Elevation Myocardial Infarction: Ischemic postconditioning or deferred stent implantation versus conventional primary angioplasty and complete revascularization versus treatment of culprit lesion only: Rationale and design of the DANAMI 3 trial program. Am Heart J. 2015 May;169(5):613-21. doi: 10.1016/j.ahj.2015.02.004. Epub 2015 Feb 14. PMID 25965708